CLINICAL TRIAL: NCT01824576
Title: Physiological Effects of Intrathoracic Pressure Regulation in Patients With Decreased Cerebral Perfusion Due to Brain Injury or Intracranial Pathology
Brief Title: Effect of Intrathoracic Pressure Regulation on Decreased Cerebral Perfusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was slower than anticipated.
Sponsor: Advanced Circulatory Systems (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACSI 5R44NS054372; 5R44NS054372 (NIH)
Record Dates: First submitted 2013-03-29; First posted 2013-04-05 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Head Injury; Intracranial Pathology; Compromised Cerebral Perfusion
Keywords: ITPR; CPP; TBI; traumatic brain injury; cerebral perfusion pressure; intrathoracic pressure regulator
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ITPR (Experimental): Use of the ITPR for 120 minutes.
  Interventions: Device: ITPR

INTERVENTIONS:
Device: ITPR — Single use noninvasive device that is connected to a vacuum source and a means to deliver a positive pressure breath. The device generates negative pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure between the periods of positive pressure ventilations.
  Other Names: Intrathoracic Pressure Regulator; CirQlator

SUMMARY:
The purpose of the study is to evaluate the physiological response to application of the Intrathoracic Pressure Regulator (ITPR) in patients with compromised cerebral circulation. The study will evaluate the physiological response to intrathoracic pressure regulation (IPR) therapy in hemodynamically stable patients with compromised cerebral circulation who are on ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* intubated and mechanically ventilated on a volume controlled mode
* head injury or other intracranial pathology and compromised cerebral perfusion
* arterial line in place or alternative with continuous pressure monitoring
* SpO2 ≥90%
* mean arterial pressure >55
* admission to ICU or about to undergo neurosurgery with planned placement of an invasive intracranial pressure monitor
* inclusion presents no significant delays to planned emergent neurosurgery
* prior written informed consent

Exclusion Criteria:

* cardiac or pulmonary injury
* confirmed pneumothorax or hemothorax
* serious neck injury resulting in neck swelling with jugular venous compression
* evidence of ongoing uncontrolled bleeding
* respiratory disease such as COPD, interstitial lung disease, or other parenchymal or pulmonary vascular disease
* marked hypertension at time of device use defined as systolic blood pressure >180 mmHg
* congestive heart failure
* women with positive serum or urine pregnancy test or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Denver, Denver, Colorado
  - Baltimore, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ITPR
Started | 9
Completed | 7
Not Completed | 2
Not completed — Device deficiency | 2

BASELINE CHARACTERISTICS:
Arm/Group | ITPR
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Black | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cerebral Perfusion Pressure (CPP)
Description: Change from average baseline CPP compared with the average CPP during use of the ITPR.
Time Frame: During 120 minutes of device use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 7
mmHg | 0.0 (6.4)

2. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: Measure change in systolic blood pressure average during baseline and 15 minutes following removal of the ITPR
Time Frame: baseline to15 minutes following device use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 7
mmHg | 9.4 (18.5)

3. Secondary Outcome: Change From Baseline in PaCO2
Description: PaCO2 will be collected during baseline and 15 minutes after device activation and change will be evaluated.
Time Frame: baseline and 15 minutes after device activation
Population: PaCO2 values for comparison were not available for two subjects
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 5
mmHg | -2.7 (3.7)

4. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Description: Measure change in diastolic blood pressure average during baseline and 15 minutes following removal of the ITPR
Time Frame: baseline to 15 minutes following device use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 7
mmHg | 4.5 (6.3)

5. Secondary Outcome: Change From Baseline in Mean Arterial Pressure (MAP)
Description: Measure change in mean arterial pressure average during baseline and 15 minutes following removal of the ITPR
Time Frame: baseline to 15 minutes following device use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 7
mmHg | 2.9 (12.9)

6. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: Measure change in heart rate average during baseline and 15 minutes following removal of the ITPR
Time Frame: baseline to 15 minutes following device use
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | ITPR
Number analyzed (Participants) | 7
beats/min | 0.3 (6.0)

7. Secondary Outcome: Change From Baseline in Pulse Pressure (PP)
Description: Measure change in pulse pressure average during baseline and 15 minutes following removal of the ITPR
Time Frame: baseline to 15 minutes following device use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 7
mmHg | 4.9 (14.8)

8. Secondary Outcome: Change From Baseline in End-tidal Carbon Dioxide (EtCO2)
Description: Measure change in EtCO2 average during baseline and 15 minutes following removal of the ITPR
Time Frame: baseline to 15 minutes following device use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 7
mmHg | 0.4 (1.6)

9. Secondary Outcome: Change From Baseline in Oxygen Saturation (SpO2)
Description: Measure change in SpO2 average during baseline and 15 minutes following removal of the ITPR
Time Frame: basseline to 15 minutes following device use
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | ITPR
Number analyzed (Participants) | 7
percentage of saturation | -0.5 (1.5)

ADVERSE EVENTS:
Arm/Group | ITPR
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITPR (N=9)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient had SpO2 desaturation to 89% likely the result of a brief ventilator disconnect
Device deficiency (Product Issues) | 1 (1) — device made a strange noise when it was turned on
Increased ICP (Vascular disorders) | 1 (1) — subject's ICP increased by >10mmHg without a concurrent rise in CerPP at the end of the run-in period before device was placed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No